CLINICAL TRIAL: NCT03822273
Title: Analgesic Effect of Acupuncture for Patients With Rib Fractures: a Randomized-controlled Trial
Brief Title: Analgesic Effect of Acupuncture for Patients With Rib Fractures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chun-Ting Liu, Attending doctor, Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201701455A3
Record Dates: First submitted 2018-12-10; First posted 2019-01-30 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Rib Fractures; Acute Pain; Analgesia
Keywords: Traumatic rib fractures; Acupuncture; Analgesia
MeSH Terms: conditions — Rib Fractures; Acute Pain; Agnosia

STUDY DESIGN:
Intervention Model Description: 1. Acupuncture group
  2. Laser acupuncture group
  3. Sham laser acupuncture group
Who Masked: Outcomes Assessor
Masking Description: All the patients are told that they will receive one kind of acupuncture treatment in addition to the original oral analgesics and assess the efficacy of acupuncture. The patients are randomly assigned to three groups after providing written informed consent, without being mentioned which kind of acupuncture treatment is applied as control. Patients are not blinded to TA or LA treatment, but they can be blinded to LA or SLA treatment. The outcome assessor is also blinded to the group assignments and is trained to apply the pain scales and conduct physical tests. To avoid unblinding of the assessment of outcomes, the patients are instructed not to discuss any aspect related to their treatment with the assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional acupuncture (TA) (Experimental): The subject will receive real acupuncture treatment once per day for 3 days after enrollment.
  Interventions: Procedure: Traditional acupuncture (TA)
- Laser acupuncture (LA) (Active Comparator): The subject will receive laser acupuncture treatment once per day for 3 days after enrollment.
  Interventions: Procedure: Laser acupuncture (LA)
- Sham laser acupuncture (SLA) (Placebo Comparator): The subject will receive sham laser acupuncture treatment once per day for 3 days after enrollment.
  Interventions: Procedure: Sham laser acupuncture (SLA)

INTERVENTIONS:
Procedure: Traditional acupuncture (TA) — Procedure: real acupuncture.
  Eight disposable, single use, sterilized, stainless steel needles are inserted at each session, and the bilateral LI4 (Hegu), SJ6 (Zhigou), ST36 (Zusanli) and GB34 (Yanglingquan) are used for acupuncture treatment. The acupuncture needles are to be inserted to a depth of 15-35 mm. All needles are rotated manually at least once at each session to elicit needle sensation (De qi). The needle retention time is 15 min.
  Arms: Traditional acupuncture (TA)
Procedure: Laser acupuncture (LA) — Procedure: laser acupuncture.
  Participants allocated to the LA group receive laser acupuncture treatment at the same acupoints used in acupuncture group. The laser acupuncture therapy will be performed with the gallium aluminum arsenide LaserPen (maximal power, 150 mW; wavelength, 810 nm; area of probe, 0.03 cm2; power density, 5 W/cm2; pulsed wave; and Bahr frequencies [B1: 599.5 Hz, B2: 1199 Hz, B3: 2398 Hz, B4: 4776 Hz, B5: 9552 Hz, B6: 19,104 Hz, and B7: 38,208 Hz]; RJ-Laser, Reimers & Janssen GmbH, Waldkirch, Germany). The laser will be applied to each point for 5 seconds, which delivered 0.375 J of energy at each of the acupoints: LI4 (Hegu, B3), SJ6 (Zhigou, B3), ST36 (Zusanli, B2) and GB34 (Yanglingquan, B2).
  Arms: Laser acupuncture (LA)
Procedure: Sham laser acupuncture (SLA) — Procedure: sham laser acupuncture.
  Subjects in the control group receive sham laser acupuncture treatment without any laser output. The acupuncture points, application duration, and total number of treatments were similar to those in the LA group.
  Arms: Sham laser acupuncture (SLA)

SUMMARY:
Traumatic rib fractures are common, resulting from significant forces impacting on the chest, and are associated with significant morbidity and mortality. Acute pain management in inpatients with traumatic rib fractures has been highly emphasized by practitioners. Inappropriate analgesia may cause respiratory complications, including pneumonia, atelectasis, acute respiratory distress syndrome, and prolonged hospital stay. These may be prevented or reduced by good analgesic therapy. This study is aimed to investigate the analgesic effect of acupuncture on traumatic rib fractures.

DETAILED DESCRIPTION:
This open-label, randomized controlled trial will involve 150 patients who have traumatic rib fractures. Subjects are randomly assigned to acupuncture group, laser acupuncture group or sham laser acupuncture group with a 1:1:1 ratio. The intervention will be performed on the consecutive three day after allocation. Bilateral LI4 (Hegu), SJ6 (Zhigou), ST36 (Zusanli) and GB34 (Yanglingquan) are used for each group. The traditional acupuncture group will be performed by inserting needles to a depth of 15-35 mm and last for 15 min. The laser acupuncture will be performed with the gallium aluminum arsenide LaserPen, which delivered 0.375 J of energy at each of the acupoints. Subjects in the control group underwent sham laser acupuncture treatment without any laser output. The acupuncture points, application duration, and total number of treatments were similar to those in the laser acupuncture group.

ELIGIBILITY:
Inclusion criteria

* Chest trauma
* Presence of one or more, unilateral or bilateral rib fractures diagnosed with chest X-ray
* Maximal rib pain score of more than 5 obtained using the numerical rating scale (NRS: 0-10)
* Ability to describe the sites of pain and evaluate the pain intensity accurately

Exclusion Criteria:

* Unable to describe the sites of pain and evaluate the pain intensity accurately
* There are open wounds on the sites of acupuncture points
* Severe multiple trauma or any poorly controlled diseases such as atelectasis, pneumonia, or other infectious diseases, immune system dysfunction, bleeding tendency, psychiatric disorders, and skin problems
* Receive surgical management of rib fractures

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Efficacy of pain relief | The NRS will be assessed at Day 1, Day 2 and DAY 3 pretreatment and posttreatment in the morning (8:00-10:00) and evening (15:00-17:00), respectively. Primary outcome is the change of NRS score on DAY 1 pretreatment and DAY 3 post treatment.
  Maximal pain intensity (Numerical Rating Scale; NRS: 0-10) evaluated by participants themselves during deep breathing, coughing, and turning over in bed.

SECONDARY OUTCOMES:
Sustained maximal inspiration lung volumes | The sustained maximal inspiration lung volumes will be assessed at Day 1, Day 2 and DAY 3 pretreatment and posttreatment in the morning (8:00-10:00) and evening (15:00-17:00), respectively.
  Sustained maximal inspiration lung volumes
Number of cases with pulmonary complications | Follow-up for one month
  Pulmonary complications including pneumonia, atelectasis, pleural effusion, acute respiratory distress syndrome, and respiratory failure.
Saliva cortisol level | The saliva cortisol level will be assessed at Day 1, Day 2 and DAY 3 pretreatment and posttreatment in the morning (8:00-10:00) and evening (15:00-17:00), respectively.
  Saliva cortisol level
Heart rate variation | The heart rate variation will be assessed at Day 1, Day 2 and DAY 3 pretreatment and posttreatment in the morning (8:00-10:00) and evening (15:00-17:00), respectively.
  Heart rate variation
The dose of narcotic and non-narcotic analgesics used | Record the medication use for 2 weeks after participant enrolled
  Record the use of narcotic and non narcotic analgesics based on chart reviews. Narcotic drugs include codeine, tramadol, and morphine. Non narcotic drugs include acetaminophen, ibuprofen, diclofenac, ketoprofen, mefenamic acid, and parecoxib.

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ting Liu, MD, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Derived] Liu CT, Hsieh TM, Wu BY, Huang YC, Shih CH, Hu WL, Tsai MY, Chen YH. Acupuncture Analgesia in Patients With Traumatic Rib Fractures: A Randomized-Controlled Trial. Front Med (Lausanne). 2022 May 27;9:896692. doi: 10.3389/fmed.2022.896692. eCollection 2022. PMID 35712110